CLINICAL TRIAL: NCT04170153
Title: An Open-label, Multicenter Trial of the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Profile of Tuvusertib (M1774) in Participants With Metastatic or Locally Advanced Unresectable Solid Tumors (DDRiver Solid Tumors 301)
Brief Title: Tuvusertib (M1774) in Participants With Metastatic or Locally Advanced Unresectable Solid Tumors (DDRiver Solid Tumors 301)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201924_0001; 2019-002203-18 (EudraCT Number); 2024-515848-23-00 (EU CTIS Number)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Metastatic or Locally Advanced Unresectable Solid Tumors
Keywords: Tuvusertib (M1774); ATR inhibitor; Niraparib; PARP inhibitor; Metastatic or Locally Advanced Unresectable Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — niraparib

STUDY DESIGN:
Intervention Model Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A1: Monotherapy Dose Escalation (Experimental): Participants will initially receive Tuvusertib (M1774) once daily under fasting conditions. Additional schedules may be evaluated if needed.
  Interventions: Drug: M1774
- Part A2 - Preliminary Food Effect Assessment (Experimental): Participants in the food effect assessment will receive Tuvusertib (M1774) at the dose and schedule determined as recommended dose for expansion (RDE) in Part A1. A single dose of Tuvusertib (M1774) will be administered on Day -7 under a fed (low-fat meal) or fasted condition, followed by a 1-week washout period. After completion of the scheduled food effect assessments, participants will follow the same schedule as participants in Part A1.
  Interventions: Drug: M1774
- Part A3 - Monotherapy Expansion (Experimental): Part A3 is an expansion of Part A1 where Tuvusertib (M1774) will be administered as a single agent at the RDE established in Part A1. Participants with defined loss-of-function mutation in ARID1A, ATRX and/or DAXX, and ATM will be enrolled.
  Interventions: Drug: M1774
- Part B1: Combination Therapy Dose Finding (Experimental): B1a: Participants with baseline body weight less than (<) 77 kilogram (kg) or platelets <150,000 cubic per millimeter (mm^3) will receive Niraparib once daily combined with different doses of Tuvusertib (M1774).
  B1b: Participants with baseline body weight greater than or equal to (>=) 77 kg and or platelets >= 150,000 mm^3 will receive Niraparib once daily combined with different doses of Tuvusertib (M1774) and schedule determined as recommended dose for expansion (RDE) in Part B1a.
  Interventions: Drug: M1774; Drug: Niraparib
- Part A4: Japan Dose Confirmation Monotherapy (Experimental): Starting at global RDE from Part A1, in Japan. Participants will initially receive Tuvusertib (M1774) once daily under fasting conditions. Additional schedules may be evaluated if needed.
  Interventions: Drug: M1774
- Part A5: China Dose Confirmation Monotherapy (Experimental): Starting at global RDE from Part A1, in China. Participants will initially receive Tuvusertib (M1774) once daily under fasting conditions. Additional schedules may be evaluated if needed.
  Interventions: Drug: M1774

INTERVENTIONS:
Drug: M1774 — M1774 will be administered orally throughout the study.
  Other Names: Tuvusertib
Drug: Niraparib — Niraparib will be administered orally throughout the study.
  Arms: Part B1: Combination Therapy Dose Finding

SUMMARY:
This is an open-label, Phase I, first-in-human (FIH) multicenter, clinical study conducted in multiple parts to establish the safety, tolerability and pharmacokinetic/pharmacodynamic (PK/PD) profile (with and without food) and early signs of efficacy of Tuvuseritib (M1774) as monotherapy and in combination with the poly (ADP-ribose) polymerase (PARP) inhibitor niraparib.

ELIGIBILITY:
Inclusion Criteria:

* Participants with locally advanced or metastatic disease that is refractory to standard therapy or for which no standard therapy is judged appropriate by the Investigator which may convey clinical benefit
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to (<=) 1
* Participants with clinically controlled brain metastases, which is defined as individuals with central nervous system metastases that have been treated for, are asymptomatic, and have discontinued steroids (for the treatment of brain metastases) for greater than (>) 28 days may be enrolled
* Participants with meningeal carcinomatosis are excluded
* In Part A3, measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
* Part A3: Participants with presence of loss of function mutations in the genes for ARID1A, ATRX and /or DAXX and ATM
* Contraceptive use by males or females will be consistent with local regulations on contraception methods for those participating in clinical studies
* Adequate hematological, hepatic, and renal function as defined in the protocol
* Female participants are not pregnant or breastfeeding
* Part B1:

Subpart B1a: Participants with Baseline Body weight < 77 kg or platelets <150,000 cubic per millimeter (mm^3) Subpart B1b: Participants with Baseline Body weight >= 77 kg and platelets >=150,000 mm^3 will be included

- Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with major surgery (as deemed by the Investigator) for any reason, except diagnostic biopsy, within 4 weeks of the study intervention and/or if the participant has not fully recovered from the surgery within 4 weeks of the study intervention
* Presence of toxicities due to prior anticancer therapies (example, radiotherapy, chemotherapy, immunotherapies, et cetera [etc]) that do not recover to <= Grade 1 with the exception of toxicities that do not pose a safety risk to the participant in the judgment of the Investigator (example: ongoing Grade 2 alopecia)
* Part B1 only: Uncontrolled arterial hypertension which is systolic blood pressure >140 millimeter of mercury (mmHg); Diastolic blood pressure >90mmHg
* Unstable angina, myocardial infarction, congestive heart failure >= II or a coronary revascularization procedure within 180 days of study entry. Calculated QTc average (using the Fridericia correction calculation) of > 450 msec for males and > 470 msec for females that does not resolve with correction of electrolyte abnormalities
* Participants with active and/or uncontrolled infection. The following exceptions apply:
* Participants with human immunodeficiency virus (HIV) infection are eligible if they are on effective antiretroviral therapy with undetectable viral load within 6 months, provided there is no expected drug-drug interaction
* Participants with evidence of chronic hepatitis B virus (HBV) infection are eligible if the HBV viral load is undetectable on suppressive therapy (if indicated), and if they have alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin levels < upper limit of normal (ULN), and provided there is no expected drug-drug interaction
* Participants with a history of hepatitis C virus (HCV) infection are eligible if they have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load, and if they have ALT, AST, and total bilirubin levels < ULN
* Treatment with live or live attenuated vaccine within 30 days of dosing (non-replicating vector vaccines are permitted)
* Part B1 only: participants diagnosed with hereditary diseases characterized by genetic defects of DNA repair mechanisms, including ataxia telangiectasia, Nijmegen breakage syndrome, Werner syndrome, Bloom Syndrome, Fanconi anemia, xeroderma pigmentosum, Cockayne syndrome, and trichothiodystrophy
* Any other clinical condition, uncontrolled concurrent illness, or other situation which in the Investigator's opinion would not make the participant a good candidate for the clinical study including or may potentially impact the absorption of M1774, such as (but not limiting to) significant small bowel resection or gastric surgery and exocrine pancreatic insufficiency requiring pancreatic enzyme replacement therapy
* Prohibited concomitant medication, as per Protocol
* Another investigational drug within 28 days or 5 half-lives, whichever is shorter, prior to start of administration of study intervention
* Prior use of Ataxia telangiectasia mutated and Rad3-related (ATR) inhibitor and/or Checkpoint kinase 1 (CHK1) inhibitor
* Participants who cannot comply with restrictions for medications or food
* Part B1 only: Participants with a known history of acute myeloid leukemia (AML) or myelodysplastic syndromes (MDS), and prostate cancer
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Part A1, A4 and A5: Occurrence of Dose-Limiting Toxicities (DLTs) During the DLT Observation Period | Day 1 to Day 21 of Cycle 1 (Each Cycle is of 21 days)
Part A1, A3, A4, A5 and B1: Occurrence of Treatment-emergent Adverse Events (TEAEs), Treatment-related Adverse Events (AEs) and Death According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A1, A3, A4, A5 and B1: Number of Participants With Grade 3 or Higher Laboratory Findings According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A1, A3, A4, A5 and B1: Number of Participants With Abnormalities in Vital Signs | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A1, A3, A4, A5 and B1: Number of Participants With Clinical Significant Abnormalities in Electrocardiogram (ECG) Findings | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A2: Area Under the Plasma Concentration Curve From Time Zero to 24 Hours Post Dose (AUC 0-24h) of Tuvusertib (M1774) | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Area Under the Plasma Concentration Curve From Time Zero to Infinity Post Dose (AUC 0-inf) of Tuvusertib (M1774) | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Maximum Observed Plasma Concentration (Cmax) of Tuvusertib (M1774) | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Relative Bioavailability Based on Area Under the Plasma Concentration Curve (Frel[AUC]) of Tuvusertib (M1774) Under Fed Condition as Compared to Fasting Condition | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Relative Bioavailability Based on Maximum Observed Plasma Concentration (Frel[Cmax]) of Tuvusertib (M1774) Under Fed Condition as Compared to Fasting Condition | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A3: Objective Response as Assessed by Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 2.2 years
Part B1: Occurrence of Dose-Limiting Toxicities (DLTs) During the DLT Observation Period | Day 1 to Day 28 of Cycle 1 (Each Cycle is of 28 days)
Part A1, A4, A5 and B1: To Determine the Recommended Dose Expansion (RDE) for Tuvusertib (M1774) monotherapy globally, in Japanese and in Chinese participants With Metastatic or Locally Advanced Unresectable Solid Tumors and in combination with Niraparib | Assessed up to approximately 2.2 years

SECONDARY OUTCOMES:
Part A1, A3, A4 and A5: Maximum Observed Plasma Concentration (Cmax) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Time to Reach Maximum Plasma Concentration (tmax) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Area Under the Plasma Concentration Curve From Time Zero to 24 Hours Post Dose (AUC0-24h) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Area Under Plasma Concentration-Time Curve Within One Dosing Interval (AUC0-tau) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Apparent Terminal Half-life (t1/2) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Apparent Total Body Clearance From Plasma (CL/f) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Apparent Clearance Body Clearance at Steady State Following Extravascular Administration (CLss/F) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Apparent Volume of Distribution During Terminal Phase Following Extravascular Administration (Vz/F) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Accumulation Ratio for Area Under the Plasma Concentration Concentration-Time Curve (Racc[AUC]) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Accumulation Ratio of Maximum Observed Plasma Concentration (Racc[Cmax]) of Tuvusertib (M1774) | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Dose Normalized Area Under Concentration-Time Curve Within One Dosing Interval (AUC0-tau/Dose) of M1774 | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24h/Dose) Post-Dose of M1774 | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Dose Normalized Area Under Concentration-Time Curve From Time Zero (dosing time) Extrapolated to Infinity (AUC0-inf/Dose) of M1774 | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M1774 | Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Area Under the Plasma Concentration Curve From Time Zero to 12 Hours (AUC0-12h) Post-Dose of M1774 | Cycle 1 Day 1 and Day 8: Pre-dose up to 12 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 12Hours (AUC0-12h/Dose) Post-dose of M1774 | Cycle 1 Day 1 and Day 8: Pre-dose upto 12 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Area Under the Plasma Concentration Curve From Time Zero to 10 Hours Post-dose (AUC0-10h) of M1774 | Part A1, A3, A4 and A5: Cycle 1 Day 1 and Day 8: Pre-dose up to 10 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 10 Hours (AUC0-10h/Dose) Post-dose of M1774 | Part A1, A3, A4 and A5: Cycle 1 Day 1 and Day 8: Pre-dose up to 10 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Area Under Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-t) of M1774 | Part A1, A3, A4 and A5: Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5 : Dose Normalized Area Under Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-t/Dose) of M1774 | Part A1, A3, A4 and A5: Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Renal Clearance (CLr) of M1774 | Part A1, A3, A4 and A5: Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Cumulative Amount Excreted From Time Zero to Infinity (Ae0-infinity) of M1774 | Part A1, A3, A4 and A5: Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Cumulative Amount Excreted From Time Zero to Time After Dosing (Ae0-t) of M1774 | Part A1, A3, A4 and A5: Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A1, A3, A4 and A5: Cumulative Percentage of Dose Excreted From Time Zero to Time After Dosing (Ae0-t%) of M1774 | Part A1, A3, A4 and A5: Cycle 1 Day 1 and Day 8: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Occurrence of Treatment-emergent Adverse Events (TEAEs), Treatment-related Adverse Events (AEs) and Death According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A2: Number of Participants With Grade 3 or Higher Laboratory Findings According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A2: Number of Participants With Abnormalities in Vital Signs | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A2: Number of Participants With Clinical Significant Abnormalities in Electrocardiogram (ECG) Findings | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A2: Time to Reach Maximum Plasma Concentration (tmax) Under Fed/Fasted Ratio of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Area Under Plasma Concentration-Time Curve Within One Dosing Interval (AUC0-tau) of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Apparent Terminal Half-life (t1/2) of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Apparent Total Body Clearance From Plasma (CL/f) of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Apparent Volume of Distribution During Terminal Phase Following Extravascular Administration (Vz/F) of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Dose Normalized Area Under Concentration Time Curve Within One Dosing Interval (AUC0-tau/Dose) of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24h/Dose) Post dose of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Dose Normalized Area Under Concentration-Time Curve From Time Zero (dosing time) Extrapolated to Infinity (AUC0-inf/Dose) of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M1774 | Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Cumulative Amount Excreted From Time Zero (dosing time) to Infinity (Ae0-inf) of M1774 | Cycle 1 Day -7: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Cumulative Amount Excreted From Time Zero to Time After Dosing (Ae0-t) of M1774 | Cycle 1 Day -7: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Cumulative Percentage of Dose Excreted From Time Zero to Time After Dosing (Ae0-t%) of M1774 | Cycle 1 Day -7: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Renal Clearance (CLr) of M1774 | Cycle 1 Day -7: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Dose Normalized Area Under Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-t/Dose) Under Fed/Fasted Ratio of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Area Under the Plasma Concentration Curve From Time Zero to 12 Hours (AUC0-12h) Post-Dose Under Fed/Fasted Ratio of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 12 hours post-dose (Each Cycle is of 21 days)
Part A2: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 12Hours (AUC0-12h/Dose) Post-dose Under Fed/Fasted Ratio of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 12 hours post-dose (Each Cycle is of 21 days)
Part A2: Area Under the Plasma Concentration Curve From Time Zero to 10 Hours PostDose AUC(0-10h) Under Fed/Fasted Ratio of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 10 hours post-dose (Each Cycle is of 21 days)
Part A2: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 10 Hours (AUC0-10h/Dose) Post-dose Under Fed/Fasted Ratio of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 10 hours post-dose (Each Cycle is of 21 days)
Part A2: Area Under Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-t) Under Fed/Fasted Ratio of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Apparent Clearance Body Clearance at Steady State Following Extravascular Administration (CLss/F) Under Fed/Fasted Ratio of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Accumulation Ratio for Area Under the Plasma Concentration Concentration-Time Curve (Racc[AUC]) Under Fed/Fasted Ratio of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Accumulation Ratio of Maximum Observed Plasma Concentration (Racc[Cmax]) Under Fed/Fasted Ratio of of M1774 | Part A2: Cycle 1 Day -7 and Day 1: Pre-dose up to 24 hours post-dose (Each Cycle is of 21 days)
Part A2: Number of Participants With Corrected QT (QTc) Interval | Baseline up to Day 8
Part A3: Duration of Response (DOR) According to RECIST v1.1 | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A3: Number of Participants With Clinical Benefit According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
  Participants with a clinical benefit, defined as an objective response or stable disease for at least 6 months, as determined by the Investigator through the use of RECIST version 1.1.
Part A3: Progression-Free Survival (PFS) as Assessed by Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part A3: Overall Survival (OS) | Baseline up to 30 days after the last dose of study treatment, assessed up to approximately 2.2 years
Part B1: Objective Response as Assessed by Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 2.2 years
Part B1: Maximum Observed Plasma Concentration (Cmax) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Time to Reach Maximum Plasma Concentration (tmax) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Area Under the Plasma Concentration Curve From Time Zero to 24 Hours Post Dose AUC(0-24h) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Area Under Plasma Concentration-Time Curve Within One Dosing Interval (AUC0-tau) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Apparent Terminal Half-life (t1/2) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Apparent Total Body Clearance From Plasma (CL/f) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Apparent Clearance Body Clearance at Steady State Following Extravascular Administration (CLss/F) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Apparent Volume of Distribution During Terminal Phase Following Extravascular Administration (Vz/F) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Accumulation Ratio for Area Under the Plasma Concentration Concentration-Time Curve (Racc[AUC]) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Accumulation Ratio of Maximum Observed Plasma Concentration (Racc[Cmax]) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Dose Normalized Area Under Concentration-Time Curve Within One Dosing Interval (AUC0-tau/Dose) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24h/Dose) Post-Dose of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Dose Normalized Area Under Concentration-Time Curve From Time Zero (dosing time) Extrapolated to Infinity (AUC0-inf/Dose) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Area Under the Plasma Concentration Curve From Time Zero to 12 Hours (AUC0-12h) Post-Dose of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3 (each cycle is of 28 days)
Part B1: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 12Hours (AUC0-12h/Dose) Post-dose of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3 (each cycle is of 28 days)
Part B1: Area Under the Plasma Concentration Curve From Time Zero to 10 Hours PostDose AUC(0-10h) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Dose Normalized Area Under Concentration-Time Curve From Time Zero to 10 Hours (AUC0-10h/Dose) Post-dose of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Area Under Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-t) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Dose Normalized Area Under Concentration-Time Curve From Time Zero to Last Sampling Time (AUC0-t/Dose) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Renal Clearance (CLr) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Cumulative Amount Excreted From Time Zero to Infinity (Ae0-infinity) of M1774 as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Cumulative Amount Excreted From Time Zero to Time After Dosing (Ae0-t) of Tuvusertib (M1774) as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)
Part B1: Cumulative Percentage of Dose Excreted From Time Zero to Time After Dosing (Ae0-t%) of Tuvusertib (M1774) as well as its Metabolites and Niraparib | Part B1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10 hours post-dose on Day 1and Day 8, Pre-dose on Day 15 of cycle 1; Pre-dose, 2, 4 hours post-dose pm Day 1 of Cycle 2; Pre-dose on Day 1 of cycle 3(each cycle is of 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (16):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - NEXT Oncology, Austin, Texas
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - University of Texas M. D. Anderson Cancer Center - Investigational Cancer Therapeutics, Houston, Texas
- Beijing Cancer Hospital, Beijing, China
- Japan (2):
  - National Cancer Center Hospital - Dept of Experimental Therapeutics, Chūōku
  - National Cancer Center Hospital East - Dept of Experimental Therapeutics, Kashiwa-shi
- Spain (4):
  - Hospital Clinic de Barcelona - Servicio de Oncologia, Barcelona
  - Hospital Universitari Vall d'Hebron - Oncology Dept., Barcelona
  - Centro Integral Oncologico Clara Campal - Unidad de Fase I-Oncologica, Madrid
  - Hospital Clinico Universitario de Valencia - Servicio de Hematologia y Oncologia Medica, Valencia
- United Kingdom (4):
  - Addenbrooke's Hospital - Dept of Oncology, Cambridge
  - The Christie Hospital - Dept of Oncology, Manchester
  - Northern Centre for Cancer Care - Sir Bobby Robson Cancer Trials Research Centre, Newcastle upon Tyne
  - Royal Marsden Hospital - Dept of Oncology, Sutton

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201924_0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: DDRiver website — http://www.DDRiver-trials.com